CLINICAL TRIAL: NCT00965276
Title: Levels of Phosphorylated AKT in Patients With Node-Positive Breast Cancer: Correlation With Disease-Free and Overall Survival
Brief Title: Relationship of pAKT to Survival in Patients With Node-Positive Breast Cancer
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040088; 04-C-0088; NCT00896870 (obsolete NCT alias)
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-12-14

CONDITIONS: Breast Cancer
Keywords: Adjuvant Therapy; Paclitaxel; Chemoresistance; Serine/Threonine Kinase; Cell Survival; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

SUMMARY:
This study will examine the relationship of a protein called pAKT to survival of breast cancer patients with one or more positive axillary lymph nodes. Akt plays a role in cell survival, tumor formation, and the development of drug resistance.

The study will use tumor tissue obtained from 2,000 patients enrolled in a National Surgical Adjuvant Breast and Bowel Project study that is evaluating whether adding the drug paclitaxel (Taxol (Registered Trademark)) to a treatment regimen of doxorubicin (Adriamycin (Registered Trademark)) and cyclophosphamide (Cytoxan (Registered Trademark)) improves disease-free survival and overall survival in patients with node-positive breast cancer. The current study will measure levels of pAkt in the tissues and correlate the results with clinical outcome to see if pAkt levels are associated with improved patient survival.

...

DETAILED DESCRIPTION:
Taxanes (paclitaxel and docetaxel) have emerged as the most powerful chemotherapeutics in breast cancer over the past decades. The B-28 clinical trial from the National Surgical Adjuvant Breast and Bowel Project (NSABP) assesses the efficacy of adding paclitaxel to the doxorubicin/cyclophosphamide regimen in the treatment of patients with axillary node positive breast cancer. The primary aim of B-28 is to determine whether four cycles of paclitaxel (Taxol (Registered Trademark)) (T) following four cycles of postoperative Doxorubicin (adriamycin (Registered Trademark) (A) and cyclophosphamide (C) will more effectively prolong disease-free survival (DFS) and survival (S) than four cycles of AC alone in patients with operable breast cancer who have one or more histologically positive axillary lymph nodes. The B-28 clinical trial tissue microarray consists of specimens from 2,000 cases enrolled. The tissue microarray set is an ideal platform for evaluating predictive markers of doxorubicin and/or paclitaxel response or resistance.

Akt, a serine/threonine protein kinase regulated by the phosphatidylinositol 3-kinase (PI3K), is of importance in cell survival, tumorigenesis, and recently shown, chemoresistance. It confers survival advantage to cells by transducing signals from growth factor receptors that activate PI3K. The primary aim of this study is to evaluate whether the levels of phosphorylated AKT are associated with disease-free and overall survival in patients with node-positive breast cancer treated with AC and/or AC followed by paclitaxel.

ELIGIBILITY:
* INCLUSION CRITERIA

The NSABP B-28 trial enrolled women from 1995 to 1998 with operable breast cancer with pathologically positive axillary lymph nodes.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2500 (Actual)
Dates: Start 2004-01-13; Study Completion 2010-12-14

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Yang SX, Costantino JP, Kim C, Mamounas EP, Nguyen D, Jeong JH, Wolmark N, Kidwell K, Paik S, Swain SM. Akt phosphorylation at Ser473 predicts benefit of paclitaxel chemotherapy in node-positive breast cancer. J Clin Oncol. 2010 Jun 20;28(18):2974-81. doi: 10.1200/JCO.2009.26.1602. Epub 2010 May 17. PMID 20479407